CLINICAL TRIAL: NCT00350207
Title: A 16-week Randomised, Placebo-controlled, Double-blind, Double-dummy, Parallel-group Study Comparing the Efficacy and Safety of Tiotropium Inhalation Solution Delivered by the Respimat Inhaler (2 Actuations of 2.5 Mcg Once Daily) With That of Salmeterol From the Hydrofluoroalkane Metered Dose Inhaler (2 Actuations of 25 Mcg Twice Daily) in Moderate Persistent Asthma Patients With the B16-Arg/Arg Genotype
Brief Title: Efficacy and Safety of Tiotropium and Salmeterol in Moderate Persistent Asthma Patients Homozygous for B16-Arg/Arg
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Model: Parallel | Purpose: Treatment
Other Study IDs: 205.342
Record Dates: First submitted 2006-07-07; First posted 2006-07-10 (Estimated); Results first posted 2009-11-17 (Estimated); Last update posted 2013-12-24 (Estimated); Status verified 2013-09

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Tiotropium Bromide; Salmeterol Xinafoate

INTERVENTIONS:
Drug: Tiotropium bromide
Drug: Placebo
Drug: Salmeterol xinafoate

SUMMARY:
This is a 16 week multicentre, multinational, randomised, double-blind, double-dummy, placebo-controlled, parallel group study to evaluate the long-term efficacy and safety of tiotropium compared to salmeterol in moderate persistent asthmatic (GINA step 3) patients homozygous for arginine at the 16th amino acid position of the beta-adrenergic receptor (ADRB2). Following an initial 4-week run-in period on salmeterol MDI patients will be randomised into the 16 week double-blind treatment period in which they receive either tiotropium once daily administered from the Respimat inhaler or salmeterol twice daily administered from the hydrofluoro-alkane Metered Dose Inhaler (MDI), or placebo twice daily. After the 16 week treatment period all patients will receive salmeterol MDI twice daily for four weeks.

The patients perform daily morning and evening peak flow (PEF) and Forced Expiratory Volume in the First Second (FEV1) measurements with an electronic peak flow meter throughout the study. Daily data on asthma control and use of rescue medication are recorded using an electronic diary included in the electronic peak flow meter. On study visits the Mini-Asthma Quality of Life Questionnaire (Elizabeth Juniper) is administered, pulse and blood pressure and pre-dose pulmonary function testing (FEV1 and Forced Vital Capacity) are performed.

ELIGIBILITY:
Inclusion_Criteria:

1. Patients homozygous for arginine at the 16th amino acid position of the beta2 adrenergic receptor (B16 Arg/Arg)
2. All patients must sign and date an Informed Consent Form for the study prior to participation in the trial
3. Male or female outpatients with at least 18 years of age, but not older than 65 years
4. Patients must have a documented history of asthma
5. Patients must be current non-smokers or ex-smokers with a cigarette smoking history of <10 pack-years
6. Patients must be on a maintenance treatment with inhaled corticosteroids with a total daily dose of 400 - 1000 mcg budesonide or equivalent

Exclusion_Criteria:

1. Patients with a significant disease other than asthma
2. Patients with a recent history (i.e., six months or less) of myocardial infarction
3. Patients who have been hospitalized for heart failure (New York Heart Association class III or IV) within the past year
4. Patients with any unstable or life threatening cardiac arrhythmia or cardiac arrhythmia requiring intervention or a change in drug therapy within the past year
5. Patients with malignancy for which the patient has undergone resection, radiation therapy or chemotherapy within the last five years. Patients with treated basal cell carcinoma are allowed.
6. Patients with a diagnosis of chronic obstructive pulmonary disease (COPD)
7. Patients with a history of life threatening pulmonary obstruction, or a history of cystic fibrosis or clinically evident bronchiectasis
8. Patients with known active tuberculosis
9. Patients who have undergone thoracotomy with pulmonary resection.
10. Patients who have completed a pulmonary rehabilitation program in the six weeks prior to visit 1 or patients who are currently in a pulmonary rehabilitation program that will not be maintained throughout the duration of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 388 (Actual)
Dates: Start 2006-07; Primary Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (109):
- Austria (7):
  - 205.342.43002 Boehringer Ingelheim Investigational Site, Graz
  - 205.342.43004 Boehringer Ingelheim Investigational Site, Trofaiach
  - 205.342.43001 Boehringer Ingelheim Investigational Site, Vienna
  - 205.342.43005 Boehringer Ingelheim Investigational Site, Vienna
  - 205.342.43006 Boehringer Ingelheim Investigational Site, Vienna
  - 205.342.43007 Boehringer Ingelheim Investigational Site, Vienna
  - 205.342.43003 Boehringer Ingelheim Investigational Site, Wels
- Belgium (13):
  - 205.342.32010 Boehringer Ingelheim Investigational Site, Anderlecht
  - 205.342.32005 Boehringer Ingelheim Investigational Site, Angleur
  - 205.342.32002 Boehringer Ingelheim Investigational Site, Brussels
  - 205.342.32007 Boehringer Ingelheim Investigational Site, Brussels
  - 205.342.32014 Boehringer Ingelheim Investigational Site, Brussels
  - 205.342.32001 Boehringer Ingelheim Investigational Site, Ghent
  - 205.342.32003 Boehringer Ingelheim Investigational Site, Herentals
  - 205.342.32004 Boehringer Ingelheim Investigational Site, Malmedy
  - 205.342.32012 Boehringer Ingelheim Investigational Site, Menen
  - 205.342.32006 Boehringer Ingelheim Investigational Site, Montigny-le-Tilleul
  - 205.342.32009 Boehringer Ingelheim Investigational Site, Namur
  - 205.342.32011 Boehringer Ingelheim Investigational Site, Turnhout
  - 205.342.32013 Boehringer Ingelheim Investigational Site, Yvoir
- Denmark (4):
  - 205.342.45003 Boehringer Ingelheim Investigational Site, Aalborg
  - 205.342.45001 Boehringer Ingelheim Investigational Site, Hvidovre
  - 205.342.45002 Boehringer Ingelheim Investigational Site, København NV
  - 205.342.45004 Boehringer Ingelheim Investigational Site, Odense C
- Finland (4):
  - 205.342.35803 Boehringer Ingelheim Investigational Site, Helsinki
  - 205.342.35801 Boehringer Ingelheim Investigational Site, Jyväskylä
  - 205.342.35802 Boehringer Ingelheim Investigational Site, Lahti
  - 205.342.35804 Boehringer Ingelheim Investigational Site, Tampere
- France (8):
  - 205.342.3305A Centre Hosp de la Cavale Blanche, Brest
  - 205.342.3304A Cabinet Médical, Chamalières
  - 205.342.3307A Boehringer Ingelheim Investigational Site, Chauny
  - 205.342.3301A UCP-X - Clinique Médicale, Grenoble
  - 205.342.3302A Hôpital Arnaud de Villeneuve, Montpellier
  - 205.342.3306A Mediscis, Poitiers
  - 205.342.3308A Boehringer Ingelheim Investigational Site, Saint Pierre La Réunion
  - 205.342.3308B Boehringer Ingelheim Investigational Site, Saint Pierre La Réunion
- Germany (14):
  - 205.342.49016 Boehringer Ingelheim Investigational Site, Beelitz-Heilstätten
  - 205.342.49004 Boehringer Ingelheim Investigational Site, Berlin
  - 205.342.49006 Boehringer Ingelheim Investigational Site, Berlin
  - 205.342.49013 Boehringer Ingelheim Investigational Site, Berlin
  - 205.342.49003 Boehringer Ingelheim Investigational Site, Bruchsal
  - 205.342.49009 Boehringer Ingelheim Investigational Site, Cologne
  - 205.342.49011 Boehringer Ingelheim Investigational Site, Frankfurt am Main
  - 205.342.49007 Boehringer Ingelheim Investigational Site, Kassel
  - 205.342.49010 Boehringer Ingelheim Investigational Site, Mainz
  - 205.342.49008 Boehringer Ingelheim Investigational Site, Minden
  - 205.342.49015 Boehringer Ingelheim Investigational Site, Neuruppin
  - 205.342.49012 Boehringer Ingelheim Investigational Site, Rathenow
  - 205.342.49005 Boehringer Ingelheim Investigational Site, Rüdersdorf
  - 205.342.49002 Boehringer Ingelheim Investigational Site, Weinheim
- Greece (6):
  - 205.342.30001 Boehringer Ingelheim Investigational Site, Athens
  - 205.342.30002 Boehringer Ingelheim Investigational Site, Athens
  - 205.342.30005 Boehringer Ingelheim Investigational Site, Heraklion
  - 205.342.30006 Boehringer Ingelheim Investigational Site, Kavala
  - 205.342.30004 Boehringer Ingelheim Investigational Site, Larissa
  - 205.342.30003 Boehringer Ingelheim Investigational Site, Thessaloniki
- Italy (8):
  - 205.342.39003 Azienda Ospedaliera " S. Anna", Ferrara
  - 205.342.39006 Azienda Ospedaliera Universitaria Careggi, Florence
  - 205.342.39005 Ospedale San Martino, Genova
  - 205.342.39002 Università di Modena e Reggio Emilia, Modena
  - 205.342.39010 Boehringer Ingelheim Investigational Site, Orbassano (to)
  - 205.342.39007 Policlinico San Matteo, Pavia
  - 205.342.39001 Ospedale di Cisanello, Pisa
  - 205.342.39009 Boehringer Ingelheim Investigational Site, Sesto San Giovanni (mi)
- Russia (8):
  - 205.342.07001 Boehringer Ingelheim Investigational Site, Moscow
  - 205.342.07002 Boehringer Ingelheim Investigational Site, Moscow
  - 205.342.07003 Boehringer Ingelheim Investigational Site, Moscow
  - 205.342.07004 Boehringer Ingelheim Investigational Site, Moscow
  - 205.342.07005 Boehringer Ingelheim Investigational Site, Moscow
  - 205.342.07006 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 205.342.07007 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 205.342.07008 Boehringer Ingelheim Investigational Site, Saint Petersburg
- Slovakia (8):
  - 205.342.42101 Boehringer Ingelheim Investigational Site, Banská Bystrica
  - 205.342.42102 Boehringer Ingelheim Investigational Site, Bratislava
  - 205.342.42104 Boehringer Ingelheim Investigational Site, Bratislava
  - 205.342.42105 Boehringer Ingelheim Investigational Site, Bratislava
  - 205.342.42107 Boehringer Ingelheim Investigational Site, Bratislava
  - 205.342.42103 Boehringer Ingelheim Investigational Site, Košice
  - 205.342.42106 Boehringer Ingelheim Investigational Site, Trenčín
  - 205.342.42108 Boehringer Ingelheim Investigational Site, Žilina
- South Africa (8):
  - 205.342.27002 Boehringer Ingelheim Investigational Site, Bellville
  - 205.342.27008 Boehringer Ingelheim Investigational Site, Bloemfontein
  - 205.342.27001 Boehringer Ingelheim Investigational Site, Cape Town
  - 205.342.27004 Boehringer Ingelheim Investigational Site, Cape Town
  - 205.342.27006 Boehringer Ingelheim Investigational Site, Centurion
  - 205.342.27003 Boehringer Ingelheim Investigational Site, Durban
  - 205.342.27007 Boehringer Ingelheim Investigational Site, George
  - 205.342.27005 Boehringer Ingelheim Investigational Site, Pretoria
- Spain (10):
  - 205.342.34006 Hospital Clinic i Provincial de Barcelona, Barcelona
  - 205.342.34011 Boehringer Ingelheim Investigational Site, Centelles
  - 205.342.34004 Hospital General Universitario de Guadalajara, Guadalajara
  - 205.342.34002 Hospital de Gran Canaria Dr. Negrín, Las Palmas de Gran Canaria
  - 205.342.34007 Hospital Universitari Arnau de Vilanova, Lleida
  - 205.342.34003 Hospital Universitario La Paz, Madrid
  - 205.342.34009 Hospital Universio Puerta del Hierro, Madrid
  - 205.342.34008 Hospital Universitario Marqués de Valdecilla, Santander
  - 205.342.34005 Hospital Vírgen de la Macarena, Seville
  - 205.342.34010 Hospital General Universitario de Valencia, Valencia
- Turkey (Türkiye) (6):
  - 205.342.90001 Boehringer Ingelheim Investigational Site, Ankara
  - 205.342.90006 Boehringer Ingelheim Investigational Site, Ankara
  - 205.342.90003 Boehringer Ingelheim Investigational Site, Bursa
  - 205.342.90007 Istanbul Universitesi Cerrahpasa Tip Fakultesi, Istanbul
  - 205.342.90005 Kocaeli Universitesi Tip Fakultesi, İzmit
  - 205.342.90004 Celal Bayar Universitesi Tip Fakultesi, Manisa
- United Kingdom (5):
  - 205.342.44002 Boehringer Ingelheim Investigational Site, Aylesbury
  - 205.342.44001 Boehringer Ingelheim Investigational Site, Chertsey
  - 205.342.44003 Boehringer Ingelheim Investigational Site, Greenisland
  - 205.342.44006 Boehringer Ingelheim Investigational Site, Leicester
  - 205.342.44005 Boehringer Ingelheim Investigational Site, Nottingham

REFERENCES:
- [Derived] Oba Y, Anwer S, Maduke T, Patel T, Dias S. Effectiveness and tolerability of dual and triple combination inhaler therapies compared with each other and varying doses of inhaled corticosteroids in adolescents and adults with asthma: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2022 Dec 6;12(12):CD013799. doi: 10.1002/14651858.CD013799.pub2. PMID 36472162
- [Derived] Bateman ED, Kornmann O, Schmidt P, Pivovarova A, Engel M, Fabbri LM. Tiotropium is noninferior to salmeterol in maintaining improved lung function in B16-Arg/Arg patients with asthma. J Allergy Clin Immunol. 2011 Aug;128(2):315-22. doi: 10.1016/j.jaci.2011.06.004. PMID 21807250

RESULTS

PARTICIPANT FLOW:
Groups:
- Tiotropium: Tiotropium inhalation solution, 5mcg once daily PM
- Salmeterol: Salmeterol Metered Aerosol, 50mcg twice daily
- Placebo: Matching Placebo
Period: Overall Study
Arm/Group | Tiotropium | Salmeterol | Placebo
Started | 128 | 134 | 126
Completed | 120 | 128 | 119
Not Completed | 8 | 6 | 7
Not completed — Adverse Event | 5 | 2 | 2
Not completed — Lack of Efficacy | 1 | 0 | 2
Not completed — Lost to Follow-up | 1 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 1
Not completed — Other | 1 | 3 | 1

BASELINE CHARACTERISTICS:
Population: Treated set includes all patients who were dispensed randomised study medication and were documented to have taken at least one dose of investigational treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Tiotropium | Salmeterol | Placebo | Total
Number analyzed (Participants) | 128 | 134 | 126 | 388
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.5 (12.6) | 42.3 (13.4) | 44.0 (11.9) | 43.3 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 82 | 83 | 75 | 240
  Male | 46 | 51 | 51 | 148

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean Weekly Morning Peak Expiratory Flow From Baseline to the End of the Trial
Description: Change from baseline in mean weekly morning peak expiratory flow at 16 weeks. Baseline is defined as the last week prior to the randomisation visit
Time Frame: baseline and after 16 weeks of treatment
Population: The Full analysis set (FAS) included patients who received at least one dose of randomised study medication and who had at least four patient diary records for at least one efficacy endpoint in any week after the first administration of the randomised treatment and baseline data for the corresponding efficacy endpoint.
Measure: Least Squares Mean (Standard Error); unit: L/min
Arm/Group | Tiotropium | Salmeterol | Placebo
Number analyzed (Participants) | 128 | 134 | 125
L/min | -3.93 (4.873) | -3.15 (4.64) | -24.63 (4.835)

2. Secondary Outcome: Mean Weekly Morning Peak Expiratory Flow at Week 4
Description: Mean weekly morning peak expiratory flow at week 4, pre-dose
Time Frame: After 4 weeks of treatment
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: L/min
Arm/Group | Tiotropium | Salmeterol | Placebo
Number analyzed (Participants) | 128 | 134 | 125
L/min | 360.695 (4.244) | 359.762 (4.041) | 335.515 (4.211)

3. Secondary Outcome: Mean Weekly Morning Peak Expiratory Flow at Week 8
Description: Mean weekly morning peak expiratory flow at week 8, pre-dose
Time Frame: After 8 weeks of treatment
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: L/min
Arm/Group | Tiotropium | Salmeterol | Placebo
Number analyzed (Participants) | 128 | 134 | 125
L/min | 355.42 (4.646) | 350.53 (4.424) | 330.193 (4.61)

4. Secondary Outcome: Mean Weekly Morning Peak Expiratory Flow at Week 12
Description: Mean weekly morning peak expiratory flow at week 12, pre-dose
Time Frame: After 12 weeks of treatment
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: L/min
Arm/Group | Tiotropium | Salmeterol | Placebo
Number analyzed (Participants) | 128 | 134 | 125
L/min | 359.05 (4.885) | 351.3 (4.652) | 332.808 (4.847)

5. Secondary Outcome: Mean Weekly Morning Peak Expiratory Flow at Week 16
Description: Mean weekly morning peak expiratory flow at week 16, pre-dose
Time Frame: After 16 weeks of treatment
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: L/min
Arm/Group | Tiotropium | Salmeterol | Placebo
Number analyzed (Participants) | 128 | 134 | 125
L/min | 355.619 (4.868) | 355.799 (4.636) | 334.525 (4.831)

6. Secondary Outcome: Mean Weekly Evening Peak Expiratory Flow at Week 4
Description: Mean weekly evening peak expiratory flow at week 4, pre-dose
Time Frame: After 4 weeks of treatment
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: L/min
Arm/Group | Tiotropium | Salmeterol | Placebo
Number analyzed (Participants) | 128 | 134 | 125
L/min | 374.496 (4.249) | 366.219 (4.045) | 348.344 (4.213)

7. Secondary Outcome: Mean Weekly Evening Peak Expiratory Flow at Week 8
Description: Mean weekly evening peak expiratory flow at week 8, pre-dose
Time Frame: After 8 weeks of treatment
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: L/min
Arm/Group | Tiotropium | Salmeterol | Placebo
Number analyzed (Participants) | 128 | 134 | 125
L/min | 368.758 (4.78) | 359.586 (4.551) | 345.299 (4.74)

8. Secondary Outcome: Mean Weekly Evening Peak Expiratory Flow at Week 12
Description: Mean weekly evening peak expiratory flow at week 12, pre-dose
Time Frame: After 12 weeks of treatment
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: L/min
Arm/Group | Tiotropium | Salmeterol | Placebo
Number analyzed (Participants) | 128 | 134 | 125
L/min | 366.282 (4.851) | 362.01 (4.617) | 344.291 (4.81)

9. Secondary Outcome: Mean Weekly Evening Peak Expiratory Flow at Week 16
Description: Mean weekly evening peak expiratory flow at week 16, pre-dose
Time Frame: After 16 weeks of treatment
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: L/min
Arm/Group | Tiotropium | Salmeterol | Placebo
Number analyzed (Participants) | 128 | 134 | 125
L/min | 363.657 (5.242) | 360.304 (4.99) | 340.099 (5.198)

10. Secondary Outcome: Mean Weekly Morning Forced Expiratory Volume in 1 Second at Week 4
Description: Mean weekly morning forced expiratory volume in 1 second at week 4, pre-dose
Time Frame: After 4 weeks of treatment
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: L
Arm/Group | Tiotropium | Salmeterol | Placebo
Number analyzed (Participants) | 128 | 134 | 125
L | 2.301 (0.026) | 2.316 (0.024) | 2.161 (0.025)

11. Secondary Outcome: Mean Weekly Morning Forced Expiratory Volume in 1 Second at Week 8
Description: Mean weekly morning forced expiratory volume in 1 second at week 8, pre-dose
Time Frame: After 8 weeks of treatment
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: L
Arm/Group | Tiotropium | Salmeterol | Placebo
Number analyzed (Participants) | 128 | 134 | 125
L | 2.254 (0.028) | 2.287 (0.027) | 2.164 (0.028)

12. Secondary Outcome: Mean Weekly Morning Forced Expiratory Volume in 1 Second at Week 12
Description: Mean weekly morning forced expiratory volume in 1 second at week 12, pre-dose
Time Frame: After 12 weeks of treatment
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: L
Arm/Group | Tiotropium | Salmeterol | Placebo
Number analyzed (Participants) | 128 | 134 | 125
L | 2.256 (0.03) | 2.254 (0.029) | 2.156 (0.03)

13. Secondary Outcome: Mean Weekly Morning Forced Expiratory Volume in 1 Second at Week 16
Description: Mean weekly morning forced expiratory volume in 1 second at week 16, pre-dose
Time Frame: After 16 weeks of treatment
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: L
Arm/Group | Tiotropium | Salmeterol | Placebo
Number analyzed (Participants) | 128 | 134 | 125
L | 2.3 (0.03) | 2.278 (0.028) | 2.188 (0.029)

14. Secondary Outcome: Mean Weekly Evening Forced Expiratory Volume in 1 Second at Week 4
Description: Mean weekly evening forced expiratory volume in 1 second at week 4, pre-dose
Time Frame: After 4 weeks of treatment
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: L
Arm/Group | Tiotropium | Salmeterol | Placebo
Number analyzed (Participants) | 128 | 134 | 125
L | 2.369 (0.029) | 2.318 (0.028) | 2.25 (0.029)

15. Secondary Outcome: Mean Weekly Evening Forced Expiratory Volume in 1 Second at Week 8
Description: Mean weekly evening forced expiratory volume in 1 second at week 8, pre-dose
Time Frame: After 8 weeks of treatment
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: L
Arm/Group | Tiotropium | Salmeterol | Placebo
Number analyzed (Participants) | 128 | 134 | 125
L | 2.32 (0.03) | 2.301 (0.029) | 2.239 (0.03)

16. Secondary Outcome: Mean Weekly Evening Forced Expiratory Volume in 1 Second at Week 12
Description: Mean weekly evening forced expiratory volume in 1 second at week 12, pre-dose
Time Frame: After 12 weeks of treatment
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: L
Arm/Group | Tiotropium | Salmeterol | Placebo
Number analyzed (Participants) | 128 | 134 | 125
L | 2.31 (0.032) | 2.299 (0.03) | 2.231 (0.032)

17. Secondary Outcome: Mean Weekly Evening Forced Expiratory Volume in 1 Second at Week 16
Description: Mean weekly evening forced expiratory volume in 1 second at week 16, pre-dose
Time Frame: After 16 weeks of treatment
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: L
Arm/Group | Tiotropium | Salmeterol | Placebo
Number analyzed (Participants) | 128 | 134 | 125
L | 2.343 (0.031) | 2.291 (0.029) | 2.215 (0.031)

18. Secondary Outcome: Mean Weekly Score for Asthma Control Diary Question "Did You Wake up During the Night Due to Asthma" at Week 4
Description: Unit on a scale 1-5. 1: Did not wake up, 2: Woke up once, 3: Woke up 2-5 times, 4: Woke up more than 5 times, 5: Was awake all night. 1 is the best value
Time Frame: After 4 weeks of treatment
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: Unit on a scale
Arm/Group | Tiotropium | Salmeterol | Placebo
Number analyzed (Participants) | 128 | 134 | 125
Unit on a scale | 1.267 (0.029) | 1.22 (0.027) | 1.232 (0.029)

19. Secondary Outcome: Mean Weekly Score for Asthma Control Diary Question "Did You Wake up During the Night Due to Asthma" at Week 8
Description: as for outcome 18
Time Frame: After 8 weeks of treatment
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: Unit on a scale
Arm/Group | Tiotropium | Salmeterol | Placebo
Number analyzed (Participants) | 128 | 134 | 125
Unit on a scale | 1.182 (0.027) | 1.176 (0.025) | 1.21 (0.027)

20. Secondary Outcome: Mean Weekly Score for Asthma Control Diary Question "Did You Wake up During the Night Due to Asthma" at Week 12
Description: as for outcome 18
Time Frame: After 12 weeks of treatment
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: Unit on a scale
Arm/Group | Tiotropium | Salmeterol | Placebo
Number analyzed (Participants) | 128 | 134 | 125
Unit on a scale | 1.203 (0.031) | 1.194 (0.03) | 1.224 (0.032)

21. Secondary Outcome: Mean Weekly Score for Asthma Control Diary Question "Did You Wake up During the Night Due to Asthma" at Week 16
Description: as for outcome 18
Time Frame: After 16 weeks of treatment
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: Unit on a scale
Arm/Group | Tiotropium | Salmeterol | Placebo
Number analyzed (Participants) | 128 | 134 | 125
Unit on a scale | 1.196 (0.034) | 1.135 (0.033) | 1.185 (0.034)

22. Secondary Outcome: Mean Weekly Score for Asthma Control Diary Question "How Were Your Asthma Symptoms in the Morning" at Week 4
Description: Unit on a scale 1-5. 1: No asthma symptoms, 2: Mild asthma symptoms, 3: Moderate asthma symptoms, 4: Severe asthma symptoms, 5: Very severe asthma symptoms. 1 is the best value
Time Frame: After 4 weeks of treatment
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: Unit on a scale
Arm/Group | Tiotropium | Salmeterol | Placebo
Number analyzed (Participants) | 128 | 134 | 125
Unit on a scale | 1.612 (0.041) | 1.486 (0.038) | 1.615 (0.041)

23. Secondary Outcome: Mean Weekly Score for Asthma Control Diary Question "How Were Your Asthma Symptoms This Morning" at Week 8
Description: as for outcome 22
Time Frame: After 8 weeks of treatment
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: Unit on a scale
Arm/Group | Tiotropium | Salmeterol | Placebo
Number analyzed (Participants) | 128 | 134 | 125
Unit on a scale | 1.504 (0.043) | 1.481 (0.041) | 1.613 (0.043)

24. Secondary Outcome: Mean Weekly Score for Asthma Control Diary Question "How Were Your Asthma Symptoms This Morning" at Week 12
Description: as for outcome 22
Time Frame: After 12 weeks of treatment
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: Unit on a scale
Arm/Group | Tiotropium | Salmeterol | Placebo
Number analyzed (Participants) | 128 | 134 | 125
Unit on a scale | 1.519 (0.046) | 1.436 (0.045) | 1.542 (0.047)

25. Secondary Outcome: Mean Weekly Score for Asthma Control Diary Question "How Were Your Asthma Symptoms This Morning" at Week 16
Description: as for outcome 22
Time Frame: After 16 weeks of treatment
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: Unit on a scale
Arm/Group | Tiotropium | Salmeterol | Placebo
Number analyzed (Participants) | 128 | 134 | 125
Unit on a scale | 1.536 (0.052) | 1.461 (0.051) | 1.647 (0.052)

26. Secondary Outcome: Mean Weekly Score for Asthma Control Diary Question "How Were Your Asthma Symptoms During the Day" at Week 4
Description: as for outcome 22
Time Frame: After 4 weeks of treatment
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: Unit on a scale
Arm/Group | Tiotropium | Salmeterol | Placebo
Number analyzed (Participants) | 128 | 134 | 125
Unit on a scale | 1.735 (0.045) | 1.637 (0.043) | 1.744 (0.045)

27. Secondary Outcome: Mean Weekly Score for Asthma Control Diary Question "How Were Your Asthma Symptoms During the Day" at Week 8
Description: as for outcome 22
Time Frame: After 8 weeks of treatment
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: Unit on a scale
Arm/Group | Tiotropium | Salmeterol | Placebo
Number analyzed (Participants) | 128 | 134 | 125
Unit on a scale | 1.603 (0.046) | 1.569 (0.043) | 1.699 (0.046)

28. Secondary Outcome: Mean Weekly Score for Asthma Control Diary Question "How Were Your Asthma Symptoms During the Day" at Week 12
Description: as for outcome 22
Time Frame: After 12 weeks of treatment
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: Unit on a scale
Arm/Group | Tiotropium | Salmeterol | Placebo
Number analyzed (Participants) | 128 | 134 | 125
Unit on a scale | 1.572 (0.05) | 1.495 (0.049) | 1.682 (0.051)

29. Secondary Outcome: Mean Weekly Score for Asthma Control Diary Question "How Were Your Asthma Symptoms During the Day" at Week 16
Description: as for outcome 22
Time Frame: After 16 weeks of treatment
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: Unit on a scale
Arm/Group | Tiotropium | Salmeterol | Placebo
Number analyzed (Participants) | 128 | 134 | 125
Unit on a scale | 1.609 (0.054) | 1.476 (0.053) | 1.711 (0.054)

30. Secondary Outcome: Mean Weekly Score for Asthma Control Diary Question "How Limited Were You in Your Activities Today Because of Your Asthma" at Week 4
Description: Unit on a scale 1-5. 1: Not limited at all, 2: A little limited, 3: Moderately limited, 4: Severely limited, 5: Totally limited. 1 is the best value
Time Frame: After 4 weeks of treatment
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: Unit on a scale
Arm/Group | Tiotropium | Salmeterol | Placebo
Number analyzed (Participants) | 128 | 134 | 125
Unit on a scale | 1.549 (0.041) | 1.514 (0.039) | 1.583 (0.041)

31. Secondary Outcome: Mean Weekly Score for Asthma Control Diary Question "How Limited Were You in Your Activities Today Because of Your Asthma" at Week 8
Description: as for outcome 30
Time Frame: After 8 weeks of treatment
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: Unit on a scale
Arm/Group | Tiotropium | Salmeterol | Placebo
Number analyzed (Participants) | 128 | 134 | 125
Unit on a scale | 1.475 (0.041) | 1.478 (0.039) | 1.545 (0.042)

32. Secondary Outcome: Mean Weekly Score for Asthma Control Diary Question "How Limited Were You in Your Activities Today Because of Your Asthma" at Week 12
Description: as for outcome 30
Time Frame: After 12 weeks of treatment
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: Unit on a scale
Arm/Group | Tiotropium | Salmeterol | Placebo
Number analyzed (Participants) | 128 | 134 | 125
Unit on a scale | 1.458 (0.045) | 1.436 (0.044) | 1.52 (0.046)

33. Secondary Outcome: Mean Weekly Score for Asthma Control Diary Question "How Limited Were You in Your Activities Today Because of Your Asthma" at Week 16
Description: as for outcome 30
Time Frame: After 16 weeks of treatment
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: Unit on a scale
Arm/Group | Tiotropium | Salmeterol | Placebo
Number analyzed (Participants) | 128 | 134 | 125
Unit on a scale | 1.446 (0.049) | 1.415 (0.047) | 1.593 (0.049)

34. Secondary Outcome: Mean Weekly Score for Asthma Control Diary Question "How Much Shortness of Breath Did You Experience During the Day" at Week 4
Description: Unit on a scale 1-5. 1: None, 2: A very little, 3: A moderate amount, 4: Quite a lot, 5: A very great deal. 1 is the best value
Time Frame: After 4 weeks of treatment
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: Unit on a scale
Arm/Group | Tiotropium | Salmeterol | Placebo
Number analyzed (Participants) | 128 | 134 | 125
Unit on a scale | 1.699 (0.045) | 1.627 (0.043) | 1.735 (0.045)

35. Secondary Outcome: Mean Weekly Score for Asthma Control Diary Question "How Much Shortness of Breath Did You Experience During the Day" at Week 8
Description: as for outcome 34
Time Frame: After 8 weeks of treatment
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: Unit on a scale
Arm/Group | Tiotropium | Salmeterol | Placebo
Number analyzed (Participants) | 128 | 134 | 125
Unit on a scale | 1.557 (0.047) | 1.571 (0.045) | 1.643 (0.048)

36. Secondary Outcome: Mean Weekly Score for Asthma Control Diary Question "How Much Shortness of Breath Did You Experience During the Day" at Week 12
Description: as for outcome 34
Time Frame: After 12 weeks of treatment
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: Unit on a scale
Arm/Group | Tiotropium | Salmeterol | Placebo
Number analyzed (Participants) | 128 | 134 | 125
Unit on a scale | 1.57 (0.048) | 1.482 (0.047) | 1.62 (0.049)

37. Secondary Outcome: Mean Weekly Score for Asthma Control Diary Question "How Much Shortness of Breath Did You Experience During the Day" at Week 16
Description: as for outcome 34
Time Frame: After 16 weeks of treatment
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: Unit on a scale
Arm/Group | Tiotropium | Salmeterol | Placebo
Number analyzed (Participants) | 128 | 134 | 125
Unit on a scale | 1.623 (0.057) | 1.482 (0.055) | 1.691 (0.057)

38. Secondary Outcome: Mean Weekly Score for Asthma Control Diary Question "Did You Experience Wheeze or Cough During the Day" at Week 4
Description: Unit on a scale 1-5. 1: Not at all, 2: A little of the time, 3: A moderate amount of the time, 4: Most of the time, 5: All the time. 1 is the best value
Time Frame: After 4 weeks of treatment
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: Unit on a scale
Arm/Group | Tiotropium | Salmeterol | Placebo
Number analyzed (Participants) | 128 | 134 | 125
Unit on a scale | 1.679 (0.048) | 1.605 (0.046) | 1.652 (0.049)

39. Secondary Outcome: Mean Weekly Score for Asthma Control Diary Question "Did You Experience Wheeze or Cough During the Day" at Week 8
Description: as for outcome 38
Time Frame: After 8 weeks of treatment
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: Unit on a scale
Arm/Group | Tiotropium | Salmeterol | Placebo
Number analyzed (Participants) | 128 | 134 | 125
Unit on a scale | 1.519 (0.05) | 1.56 (0.047) | 1.575 (0.05)

40. Secondary Outcome: Mean Weekly Score for Asthma Control Diary Question "Did You Experience Wheeze or Cough During the Day" at Week 12
Description: as for outcome 38
Time Frame: After 12 weeks of treatment
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: Unit on a scale
Arm/Group | Tiotropium | Salmeterol | Placebo
Number analyzed (Participants) | 128 | 134 | 125
Unit on a scale | 1.539 (0.051) | 1.505 (0.05) | 1.572 (0.052)

41. Secondary Outcome: Mean Weekly Score for Asthma Control Diary Question "Did You Experience Wheeze or Cough During the Day" at Week 16
Description: as for outcome 38
Time Frame: After 16 weeks of treatment
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: Unit on a scale
Arm/Group | Tiotropium | Salmeterol | Placebo
Number analyzed (Participants) | 128 | 134 | 125
Unit on a scale | 1.528 (0.057) | 1.515 (0.056) | 1.669 (0.057)

42. Secondary Outcome: Morning Pre-dose Forced Expiratory Volume in 1 Second as Measured by Spirometry at Visit 3
Description: Morning pre-dose forced expiratory volume in 1 second as measured by spirometry after 6 weeks of treatment
Time Frame: After 6 weeks of treatment
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: L
Arm/Group | Tiotropium | Salmeterol | Placebo
Number analyzed (Participants) | 128 | 134 | 125
L | 2.471 (0.031) | 2.401 (0.03) | 2.299 (0.031)

43. Secondary Outcome: Morning Pre-dose Forced Expiratory Volume in 1 Second as Measured by Spirometry at Visit 4
Description: Morning pre-dose forced expiratory volume in 1 second as measured by spirometry after 12 weeks of treatment
Time Frame: After 12 weeks of treatment
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: L
Arm/Group | Tiotropium | Salmeterol | Placebo
Number analyzed (Participants) | 128 | 134 | 125
L | 2.467 (0.031) | 2.442 (0.03) | 2.266 (0.031)

44. Secondary Outcome: Morning Pre-dose Forced Expiratory Volume in 1 Second as Measured by Spirometry at Visit 5
Description: Morning pre-dose forced expiratory volume in 1 second as measured by spirometry after 16 weeks od treatment
Time Frame: After 16 weeks of treatment
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: L
Arm/Group | Tiotropium | Salmeterol | Placebo
Number analyzed (Participants) | 128 | 134 | 125
L | 2.439 (0.03) | 2.457 (0.029) | 2.29 (0.03)

45. Secondary Outcome: Morning Pre-dose Forced Vital Capacity as Measured by Spirometry at Visit 3
Description: Morning pre-dose forced vital capacity as measured by spirometry after 6 weeks of treatment
Time Frame: After 6 weeks of treatment
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: L
Arm/Group | Tiotropium | Salmeterol | Placebo
Number analyzed (Participants) | 128 | 134 | 125
L | 3.531 (0.034) | 3.441 (0.033) | 3.367 (0.034)

46. Secondary Outcome: Morning Pre-dose Forced Vital Capacity as Measured by Spirometry at Visit 4
Description: Morning pre-dose forced vital capacity as measured by spirometry after 12 weeks of treatment
Time Frame: After 12 weeks of treatment
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: L
Arm/Group | Tiotropium | Salmeterol | Placebo
Number analyzed (Participants) | 128 | 134 | 125
L | 3.509 (0.035) | 3.495 (0.033) | 3.307 (0.034)

47. Secondary Outcome: Morning Pre-dose Forced Vital Capacity as Measured by Spirometry at Visit 5
Description: Morning pre-dose forced vital capacity as measured by spirometry after 16 weeks of treatment
Time Frame: After 16 weeks of treatment
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: L
Arm/Group | Tiotropium | Salmeterol | Placebo
Number analyzed (Participants) | 128 | 134 | 125
L | 3.488 (0.034) | 3.474 (0.033) | 3.353 (0.034)

48. Secondary Outcome: Mini-Asthma Quality of Life Questionnaire (Mini-AQLQ) Overall Score at Visit 3
Description: Mean of the responses to 15 questions from 4 domains: Symptoms (1), Activity Limitations (2), Emotional Function (3), Environmental Stimuli (4). Unit on a scale 1-7. For domain (2): 1: totally limited, 2: extremely limited, 3: very limited, 4: moderate limitation, 5: some limitation, 6: a little limitation, 7: not at all limited. For other domains: 1: all of the time, 2: most of the time, 3: a good bit of the time, 4: some of the time, 5: a little of the time, 6: hardly any of the time, 7: none of the time. 7 is the best value
Time Frame: After 6 weeks of treatment
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: Unit on a scale
Arm/Group | Tiotropium | Salmeterol | Placebo
Number analyzed (Participants) | 128 | 134 | 125
Unit on a scale | 5.050 (0.067) | 5.259 (0.064) | 5.097 (0.067)

49. Secondary Outcome: Mini-AQLQ Overall Score at Visit 4
Description: as for outcome 48
Time Frame: After 12 weeks of treatment
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: Unit on a scale
Arm/Group | Tiotropium | Salmeterol | Placebo
Number analyzed (Participants) | 128 | 134 | 125
Unit on a scale | 5.233 (0.066) | 5.399 (0.063) | 5.078 (0.066)

50. Secondary Outcome: Mini-AQLQ Overall Score at Visit 5
Description: as for outcome 48
Time Frame: After 16 weeks of treatment
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: Unit on a scale
Arm/Group | Tiotropium | Salmeterol | Placebo
Number analyzed (Participants) | 128 | 134 | 125
Unit on a scale | 5.305 (0.068) | 5.454 (0.064) | 5.214 (0.067)

51. Secondary Outcome: Systolic Blood Pressure in Conjunction With Spirometry at Visit 3
Description: Systolic blood pressure collected in conjunction with spirometry at 6 weeks
Time Frame: After 6 weeks of treatment
Population: Treated set. Some patients discontinued the trial between Visits. Thus these patients are in the efficacy analysis for the respective period (are added in the participant flow) but they have no safety blood pressure/pulse rate measurements, because blood pressure and pulse rate were measured at Visits
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Tiotropium | Salmeterol | Placebo
Number analyzed (Participants) | 126 | 131 | 122
mmHg | 124.68 (14.53) | 123.11 (11.5) | 126.41 (14.48)

52. Secondary Outcome: Systolic Blood Pressure in Conjunction With Spirometry at Visit 4
Description: Systolic blood pressure collected in conjunction with spirometry at 12 weeks
Time Frame: After 12 weeks of treatment
Population: as for outcome 51
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Tiotropium | Salmeterol | Placebo
Number analyzed (Participants) | 121 | 129 | 119
mmHg | 124.81 (13.86) | 123.92 (12.15) | 125.18 (13.45)

53. Secondary Outcome: Systolic Blood Pressure in Conjunction With Spirometry at Visit 5
Description: Systolic blood pressure collected in conjunction with spirometry at 16 weeks
Time Frame: After 16 weeks of treatment
Population: as for outcome 51
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Tiotropium | Salmeterol | Placebo
Number analyzed (Participants) | 122 | 128 | 119
mmHg | 124.23 (14.59) | 123.83 (12.82) | 124.47 (13.77)

54. Secondary Outcome: Diastolic Blood Pressure in Conjunction With Spirometry at Visit 3
Description: Diastolic blood pressure collected in conjunction with spirometry at 6 weeks
Time Frame: After 6 weeks of treatment
Population: as for outcome 51
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Tiotropium | Salmeterol | Placebo
Number analyzed (Participants) | 126 | 131 | 122
mmHg | 78.62 (9.26) | 77.62 (8.74) | 79.34 (8.37)

55. Secondary Outcome: Diastolic Blood Pressure in Conjunction With Spirometry at Visit 4
Description: Diastolic blood pressure collected in conjunction with spirometry at 12 weeks
Time Frame: After 12 weeks of treatment
Population: as for outcome 51
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Tiotropium | Salmeterol | Placebo
Number analyzed (Participants) | 121 | 129 | 119
mmHg | 77.88 (9.93) | 77.22 (9.23) | 78.29 (8.04)

56. Secondary Outcome: Diastolic Blood Pressure in Conjunction With Spirometry at Visit 5
Description: Diastolic blood pressure collected in conjunction with spirometry at 16 weeks
Time Frame: After 16 weeks of treatment
Population: as for outcome 51
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Tiotropium | Salmeterol | Placebo
Number analyzed (Participants) | 122 | 128 | 119
mmHg | 79.23 (9.35) | 77.61 (7.92) | 78.38 (9.38)

57. Secondary Outcome: Pulse Rate in Conjunction With Spirometry at Visit 3
Description: Pulse rate collected in conjunction with spirometry at 6 weeks
Time Frame: After 6 weeks of treatment
Population: as for outcome 51
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Tiotropium | Salmeterol | Placebo
Number analyzed (Participants) | 125 | 131 | 121
bpm | 74.7 (8.8) | 74.9 (8.4) | 74.2 (9.4)

58. Secondary Outcome: Pulse Rate in Conjunction With Spirometry at Visit 4
Description: Pulse rate collected in conjunction with spirometry at 12 weeks
Time Frame: After 12 weeks of treatment
Population: as for outcome 51
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Tiotropium | Salmeterol | Placebo
Number analyzed (Participants) | 121 | 129 | 119
bpm | 74.8 (9.9) | 74.6 (9.2) | 74.2 (8.4)

59. Secondary Outcome: Pulse Rate in Conjunction With Spirometry at Visit 5
Description: Pulse rate collected in conjunction with spirometry at 16 weeks
Time Frame: After 16 weeks of treatment
Population: as for outcome 51
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Tiotropium | Salmeterol | Placebo
Number analyzed (Participants) | 121 | 128 | 119
bpm | 74.4 (9.9) | 75.3 (8.3) | 74.7 (10.1)

60. Secondary Outcome: Mean PEF Variability at Week 4
Description: PEF (Peak expiratory flow) variability is defined as the difference between the highest morning PEF value and the highest evening PEF value of one day divided by the arithmetic mean of these two PEF values and multiplied by 100%
Time Frame: After 4 weeks of treatment
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: ratio expressed in percent
Arm/Group | Tiotropium | Salmeterol | Placebo
Number analyzed (Participants) | 128 | 134 | 125
ratio expressed in percent | 12.043 (0.611) | 10.547 (0.584) | 12.085 (0.606)

61. Secondary Outcome: Mean PEF Variability at Week 8
Description: as for outcome 60
Time Frame: After 8 weeks of treatment
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: ratio expressed in percent
Arm/Group | Tiotropium | Salmeterol | Placebo
Number analyzed (Participants) | 128 | 134 | 125
ratio expressed in percent | 13.377 (0.695) | 11.252 (0.664) | 12.964 (0.689)

62. Secondary Outcome: Mean PEF Variability at Week 12
Description: as for outcome 60
Time Frame: After 12 weeks of treatment
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: ratio expressed in percent
Arm/Group | Tiotropium | Salmeterol | Placebo
Number analyzed (Participants) | 128 | 134 | 125
ratio expressed in percent | 11.735 (0.654) | 11.320 (0.625) | 11.257 (0.648)

63. Secondary Outcome: Mean PEF Variability at Week 16
Description: as for outcome 60
Time Frame: After 16 weeks of treatment
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: ratio expressed in percent
Arm/Group | Tiotropium | Salmeterol | Placebo
Number analyzed (Participants) | 128 | 134 | 125
ratio expressed in percent | 11.742 (0.656) | 10.793 (0.627) | 12.305 (0.650)

ADVERSE EVENTS:
Time Frame: From first study drug administration until 30 days after last randomised study drug administration
Arm/Group | Tiotropium | Salmeterol | Placebo
Serious Adverse Events (participants affected / at risk) | 2/128 | 7/134 | 1/126
Other Adverse Events (participants affected / at risk) | 21/128 | 18/134 | 25/126
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tiotropium (N=128) | Salmeterol (N=134) | Placebo (N=126)
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0
Meningitis (Infections and infestations) | 1 | 0 | 0
Pilonidal cyst (Infections and infestations) | 1 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Ligament injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tiotropium (N=128) | Salmeterol (N=134) | Placebo (N=126)
Nasopharyngitis (Infections and infestations) | 5 | 3 | 9
Asthma (Respiratory, thoracic and mediastinal disorders) | 16 | 15 | 16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.